CLINICAL TRIAL: NCT06930807
Title: Development and Validation of Non-Invasive Monitoring Techniques for Postoperative Recurrence and Novel Adjuvant Therapeutic Strategies in Lung Cancer
Brief Title: Liquid Biopsy-Based Novel Modality for Postoperative Management of Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other); Guangdong Provincial People's Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Shanghai Chest Hospital (Other); Shandong Cancer Hospital and Institute (Other); Shenzhen Third People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Shanghai Zhongshan Hospital (Other); Peking University First Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chen KeZhong, Professor, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0501900
Record Dates: First submitted 2025-03-25; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer; Minimal Residual Disease; Adaptive Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adaptive postoperative management group (Experimental): For those who don't receive neoadjuvant therapy, if the MRD testing results after surgery keep negative, postoperative adjuvant therapy will be waived.
  For those who receive neoadjuvant therapy, if the efficacy reaches pathological complete response(pCR) and MRD testing results keep negative, postoperative adjuvant therapy will be waived.
  Otherwise, participants will receive a customized treatment plan based on Multi-disciplinary Treatment (MDT).
  Interventions: Other: Adaptive postoperative management based on minimal residual disease
- standard clinical postoperative management group (No Intervention): These participants will receive standard postoperative adjuvant therapy and routine follow-up.

INTERVENTIONS:
Other: Adaptive postoperative management based on minimal residual disease — participants will not receive postoperative treatment if (neoadjuvant therapy efficacy reaches pCR and) MRD results keep negative.
  Arms: adaptive postoperative management group

SUMMARY:
The goal of this study is to develop new techniques for minimal residual disease(MRD) monitoring and to confirm the efficacy and safety of MRD-guided postoperative management for early stage non-small cell lung cancer. The main questions this study aims to answer are:

* How to develop multi-omics-based high-sensitivity detection methods to accurately capture MRD and monitor postoperative recurrence in lung cancer?
* Is adaptive treatment guided by ctDNA-MRD for lung cancer patients superior to traditional clinical management and effectively improves survival?
* Do heterogeneous patient populations (grouped by stages, histopathological subtypes, driver mutations, and treatment histories) show differences in effects under ctDNA-MRD guided postoperative management strategies?

DETAILED DESCRIPTION:
Approximately 30% of early-stage lung cancer patients experience recurrence after curative surgery. However, the clinical utility of routine chest CT surveillance remains limited. Emerging evidence has demonstrated that liquid biopsy-based minimal residual disease (MRD) detection may serve as a more sensitive monitoring strategy. Longitudinal ctDNA dynamics analysis further enables real-time assessment of tumor progression and early detection of molecular relapse.

This study aims to develop a novel multidimensional approach for non-invasive postoperative recurrence monitoring in lung cancer and establish an MRD-guided adjuvant therapy model to optimize precision treatment and MRD-stratified follow-up protocols for lung cancer patients. This study will evaluate the sensitivity and specificity of novel monitoring methods and further compare emerging non-invasive recurrence monitoring approaches with conventional ctDNA-based techniques, driving continuous advancements in lung cancer research.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer with stage IA-IIIA (8th edition TNM classification) planning to undergo curative surgery or to undergo neoadjuvant therapy
* Solid nodules >1 cm or ground-glass nodules >1.5 cm on imaging
* No history of malignancies other than non-small cell lung cancer in the past 5 years
* Specimens are well preserved and imaging documents are accessible.

Exclusion Criteria:

* Age<18 years old
* Non-small cell lung cancer with pathologic stage IIIB-IV (8th edition TNM classification)
* Pathology results confirmed not to be non-small cell lung cancer
* History of malignancies other than non-small cell lung cancer in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Two-year recurrence-free survival rate | Time from curative surgery to confirmation of clinical progression (recurrence or metastasis) within two years.
  The difference in the proportion of patients with (suspected) relapse or metastasis between the intervention group and the control group within two years.

SECONDARY OUTCOMES:
Overall survival | Time from curative surgery to confirmation of death (any cause)，assessed up to 60 months.
  The difference in overall survival between the intervention group and the control group.
Incremental cost effectiveness ratio | 24 months after surgery
  The cost of lung cancer-related treatment, including the cost of drugs, follow-up treatment, drug management costs (consultation fees, anti-tumor drug allocation fees, intravenous infusion fees, nursing fees, etc.), follow-up costs, laboratory tests and imaging examination costs, and the management costs of adverse reactions (1 cycle is counted as 1 time), and the per capita standard expenses calculated according to the Checkmate816 study protocol and China's expenses were used to calculate ICER.
Timely diagnosis rate by the novel MRD monitoring technique | two years
  The proportion of patients with recurrence signals detected by non-invasive methods prior to clinical confirmation of recurrence/metastasis, and quantify the mean lead time.
Sensitivity of the novel MRD monitoring approach | two years
  Evaluate the sensitivity of the novel MRD-based assay against previous ctDNA-MRD-only approaches. Use receiver operating characteristic (ROC) curves and limit of detection (LoD) analyses for cross-platform comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Chen, MD, Study Chair — Peking University People's Hospital; Guangxi Wang, PhD, Study Director — Peking University; Jiatao Zhang, MD, Study Director — Guangdong Provincial People's Hospital; Rong Yin, MD, Study Director — Jiangsu Cancer Institute & Hospital; Ziming Li, MD, Study Director — Shanghai Chest Hospital; Yintao Li, MD, Principal Investigator — Shandong Cancer Hospital and Institute; Zizi Zhou, MD, Principal Investigator — Shenzhen Third People's Hospital; Fang Wu, MD, Principal Investigator — Second Xiangya Hospital of Central South University; Jun Yin, MD, Principal Investigator — Shanghai Zhongshan Hospital; Yuan Cheng, MD, Principal Investigator — Peking University First Hospital; Quanfu Huang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Xiaojun Zhu, PhD, Principal Investigator — China National Institute for Occupational Safety and Health (NIOSH/CDC)
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided